CLINICAL TRIAL: NCT04435938
Title: A Phase 2 Study of SBRT for Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of SBRT for Squamous Cell Carcinoma of the Head and Neck
Acronym: SHINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8134
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-06

CONDITIONS: Head and Neck Neoplasms; Squamous Cell Carcinoma; Squamous Skin Carcinoma
Keywords: Head and Neck Cancer; Squamous Cell Cancer; Squamous Skin Cancer; Stereotactic Body Radiotherapy; SBRT; Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Eligible and consenting patients will be treated with the dose prescribed in the study of 45Gy in 5 fractions, delivered once every 3-4 days, such that treatment is completed within 15 days (Exceptions: treatment duration of up to 18 days will be allowed to account for cancer centre closures and unforeseen patient issues). Using the Simon optimal two-stage design, 11 patients will be recruited in the first stage. If 6 or less patients have a response, the study will be stopped at the end of stage I, however, if 7 or more patients have a response the study will continue to stage II, in which an additional 27 patients (for a total of 38) will be recruited. At the end of stage II, if 26 or less patients have a response, then H0 will be accepted and the treatment regimen deemed not worthy of further study, however, if 27 or more patients have a response, the treatment regimen will be recommended for further study in phase III.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): The dose prescribed in the study will be 45Gy in 5 fractions, delivered once every 3-4 days, such that treatment is completed within 15 days. (e.g. treatment given on Monday/Thursday/Mon/Thurs/Mon) (Exceptions: treatment duration of up to 18 days will be allowed to account for cancer centre closures and unforeseen patient issues.)
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — 45 Gy in 5 fractions delivered once every 3-4 days

SUMMARY:
To evaluate the tumour response rate of squamous cell carcinoma of the head and neck following stereotactic body radiotherapy (SBRT) of 45Gy in 5 fractions delivered once every 3-4 days, such that treatment is completed within 15 days.

DETAILED DESCRIPTION:
Cancers of the head and neck region account for approximately 4% of all new cancer cases. Primary skin cancers are the most common malignancy diagnosed in North America with the majority of tumours arising in the cervico-facial region.Together, these tumours comprise a high burden of illness and are often characterized by locally advanced, non-metastatic disease.

Determining the optimal treatment for individual patients with advanced cervico-facial cancers of the skin or primary head and neck squamous cell carcinoma (HNSCC) is clinically challenging; standard treatments include combinations of surgery, radiation and chemotherapy, all of which are associated with high rates of acute toxicity and complications. A meta-analysis of randomized controlled trials did not demonstrate benefit with concurrent chemotherapy in patients over the age of 70 or with performance status ≥ 2, and it is recognized that the high burden of medical co-morbidities in HNSCC is associated with poorer prognosis. Some patients without distant metastases may be deemed to have 'incurable' disease due to very advanced tumours, recurrence, severe medical co-morbidities or frailty that prohibit the use of standard surgery, general anaesthetic and/or radiotherapy over 6-7 weeks.

When conventional surgery and/or radiotherapy are not recommended by the multi-disciplinary team then patients may be treated with shorter, hypo-fractionated radiotherapy with the goal of symptom relief and local control but at the cost of a lower biological dose. Investigators at the Juravinski Cancer Centre published retrospective results from the '0-7-21' regimen using 24 Gy / 3 fractions which was well tolerated and provided temporary symptom relief in 82% of patients but reported 6 month progression free survival of 39% within the irradiated field; a phase 2 study of previously untreated HNSCC patients deemed to have incurable disease used up to 42 Gy/12 fractions and demonstrated similar rates of initial response and symptom relief but a short progression free survival duration of 3.1 months. One study reported an institutional experience of palliative radiotherapy in newly diagnosed head and neck cancer patients who were deemed to have incurable disease and received a wide range of dose/fractionation regimens. The median radiation dose was 50 Gy and between 57-82% of patients were reported to have any radiological, clinical or symptomatic response to treatment. In these three studies, the patients were older with median ages of 71, 73, and 77 years - and median survival was short 5.2, 5.7 and 6.2 months.

With respect to squamous cell carcinoma (SCC) of the skin, there is limited evidence to guide treatment in patients with unresectable or medically inoperable disease, particularly in the head and neck region. There is a need for prospective data on non-surgical treatment options for frail older adults which improve efficacy while limiting the treatment burden.

SBRT can limit the number of treatments while delivering a higher, potentially curative dose. An international consortium of 15 high volume cancer centres reported on a survey of practices using SBRT for head and neck cancers. There was heterogeneity in the indications, techniques and doses reported by various institutions. The most common indication was in the setting of recurrent disease and reported doses were in the range of 35-50 Gy in 3-5 fractions. Several institutions reported 1-2 year local control rates of 65-90% with SBRT and acceptable levels of toxicity. To our knowledge, there are no prospective clinical studies evaluating tumour response, toxicity and quality of life in previously unirradiated patients.

The goal of the current study is to prospectively evaluate tumour response, toxicity and patient quality of life in patients with HNSCC undergoing SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 60 years
2. Histologically confirmed diagnosis of squamous cell carcinoma of the head and neck region including primary skin SCC; (malignant cells with suspicious/likely SCC will be considered for study if repeat biopsy is not feasible)
3. Clinical stage ≥ T2, or any T-stage with N1-N3 disease, M0 or Mx
4. Measurable tumour present in the head and neck region on clinical examination and/or imaging at time of study enrollment
5. All patients will be assessed by a multi-disciplinary, head and neck oncology team with no systemic therapy being recommended at the time of enrollment
6. Primary surgery not recommended/performed due to any of the following:

   * Unresectable disease and/or borderline resectable
   * Medically inoperable / deemed high risk for post-operative morbidity/mortality by surgical team
   * Patient declined surgery
7. Deemed not to be a candidate for standard fractionation radiotherapy due to poor performance status and/or medical co-morbidities and/or advanced stage disease
8. Eastern Co-operative Oncology Group (ECOG) Performance Status ≤ 3

Exclusion Criteria:

1. Life expectancy ≤ 3 months
2. Chemotherapy or other systemic cancer therapy within 3 months prior to HN SBRT
3. Basal cell carcinoma, Merkel cell, malignant melanoma, adenocarcinoma are excluded
4. HN surgery within 6 months prior to HN SBRT (excision under local anaesthesia is acceptable)
5. Prior radiation treatment to the head and neck region (prior radiotherapy to the skin for non-melanoma skin cancer and deemed to have no risk of overlap with the current field are eligible)
6. Synchronous or recent cancer diagnosis not including the index cancer (other cancers treated curatively with no evidence of disease for >=3 years, or other non- melanoma skin cancers treated with no evidence of disease for >= 6 months are eligible)
7. Confirmed or known distant metastatic disease.
8. Serious non-malignant disease that precludes definitive radiation treatment (e.g.

   severe cases of scleroderma, systemic lupus erythematosus, rheumatoid arthritis)
9. Unable to provide written, informed consent or complete QoL questionnaires and assessments required on the study
10. Unable to lie flat for 60 minutes in order to have radiation planning and treatment
11. Unable to attend radiation planning and therapy, as well as follow-up care and assessments
12. Unable to provide written, informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Tumour response rate | The best overall response across all time points during the study period - up to 24 months after completion of SBRT.
  Tumour response rate defined as complete or partial response according to Tumour response rate will be defined by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Number of participants with Acute and Late Toxicity | Up to 24 months after completion of SBRT
  Acute toxicity (during and up to 3 months from the end of treatment) and late toxicity (after 3 months) adverse effects secondary to SBRT treatment will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0) scale.
Local Control | Determination of local recurrence will be based on based on RECIST criteria 1.1 (see section 11.3 below) and assessed on MRI or CT scan imaging at 12 weeks and any additional imaging/clinical assessments performed during the study.
  The absence of local progression of disease of the target lesions during the study period.
Quality of Life as measured by the FACT-HN questionnaire | The FACT-HN Quesionnaire will be administered at Baseline, once during treatment, 6 weeks, 3, 6, 12 months post SBRT treatment. Higher scores represent better qualtiy of life.
  Assessed using the FACT-HN questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lee, MD, Principal Investigator — Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Eskander A, Krzyzanowska MK, Fischer HD, Liu N, Austin PC, Irish JC, Enepekides DJ, Lee J, Gutierrez E, Lockhart E, Raphael M, Singh S. Emergency department visits and unplanned hospitalizations in the treatment period for head and neck cancer patients treated with curative intent: A population-based analysis. Oral Oncol. 2018 Aug;83:107-114. doi: 10.1016/j.oraloncology.2018.06.011. Epub 2018 Jun 19. PMID 30098764
- [Background] Pignon JP, le Maitre A, Maillard E, Bourhis J; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): an update on 93 randomised trials and 17,346 patients. Radiother Oncol. 2009 Jul;92(1):4-14. doi: 10.1016/j.radonc.2009.04.014. Epub 2009 May 14. PMID 19446902
- [Background] Reid BC, Alberg AJ, Klassen AC, Samet JM, Rozier RG, Garcia I, Winn DM. Comorbidity and survival of elderly head and neck carcinoma patients. Cancer. 2001 Oct 15;92(8):2109-16. doi: 10.1002/1097-0142(20011015)92:83.0.co;2-m. PMID 11596027
- [Background] Datema FR, Ferrier MB, van der Schroeff MP, Baatenburg de Jong RJ. Impact of comorbidity on short-term mortality and overall survival of head and neck cancer patients. Head Neck. 2010 Jun;32(6):728-36. doi: 10.1002/hed.21245. PMID 19827120
- [Background] Nguyen NT, Doerwald-Munoz L, Zhang H, Kim DH, Sagar S, Wright JR, Hodson DI. 0-7-21 hypofractionated palliative radiotherapy: an effective treatment for advanced head and neck cancers. Br J Radiol. 2015 May;88(1049):20140646. doi: 10.1259/bjr.20140646. Epub 2015 Feb 19. PMID 25694259
- [Background] Corry J, Peters LJ, Costa ID, Milner AD, Fawns H, Rischin D, Porceddu S. The 'QUAD SHOT'--a phase II study of palliative radiotherapy for incurable head and neck cancer. Radiother Oncol. 2005 Nov;77(2):137-42. doi: 10.1016/j.radonc.2005.10.008. Epub 2005 Nov 2. PMID 16260054
- [Background] Stevens CM, Huang SH, Fung S, Bayley AJ, Cho JB, Cummings BJ, Dawson LA, Hope AJ, Kim JJ, O'Sullivan B, Waldron JN, Ringash J. Retrospective study of palliative radiotherapy in newly diagnosed head and neck carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):958-63. doi: 10.1016/j.ijrobp.2010.06.055. Epub 2010 Oct 14. PMID 20950952
- [Background] Lansbury L, Bath-Hextall F, Perkins W, Stanton W, Leonardi-Bee J. Interventions for non-metastatic squamous cell carcinoma of the skin: systematic review and pooled analysis of observational studies. BMJ. 2013 Nov 4;347:f6153. doi: 10.1136/bmj.f6153. PMID 24191270
- [Background] Lubeek SF, Borgonjen RJ, van Vugt LJ, Olde Rikkert MG, van de Kerkhof PC, Gerritsen MJ. Improving the applicability of guidelines on nonmelanoma skin cancer in frail older adults: a multidisciplinary expert consensus and systematic review of current guidelines. Br J Dermatol. 2016 Nov;175(5):1003-1010. doi: 10.1111/bjd.14923. Epub 2016 Sep 13. PMID 27484632
- [Background] Karam I, Yao M, Heron DE, Poon I, Koyfman SA, Yom SS, Siddiqui F, Lartigau E, Cengiz M, Yamazaki H, Hara W, Phan J, Vargo JA, Lee V, Foote RL, Harter KW, Lee NY, Sahgal A, Lo SS. Survey of current practices from the International Stereotactic Body Radiotherapy Consortium (ISBRTC) for head and neck cancers. Future Oncol. 2017 Mar;13(7):603-613. doi: 10.2217/fon-2016-0403. Epub 2016 Nov 15. PMID 27842456
- [Background] Khan L, Tjong M, Raziee H, Lee J, Erler D, Chin L, Poon I. Role of stereotactic body radiotherapy for symptom control in head and neck cancer patients. Support Care Cancer. 2015 Apr;23(4):1099-103. doi: 10.1007/s00520-014-2421-y. Epub 2014 Oct 9. PMID 25294656
- [Background] Vargo JA, Ferris RL, Ohr J, Clump DA, Davis KS, Duvvuri U, Kim S, Johnson JT, Bauman JE, Gibson MK, Branstetter BF, Heron DE. A prospective phase 2 trial of reirradiation with stereotactic body radiation therapy plus cetuximab in patients with previously irradiated recurrent squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):480-8. doi: 10.1016/j.ijrobp.2014.11.023. Epub 2015 Jan 30. PMID 25680594
- [Background] Heron DE, Ferris RL, Karamouzis M, Andrade RS, Deeb EL, Burton S, Gooding WE, Branstetter BF, Mountz JM, Johnson JT, Argiris A, Grandis JR, Lai SY. Stereotactic body radiotherapy for recurrent squamous cell carcinoma of the head and neck: results of a phase I dose-escalation trial. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1493-500. doi: 10.1016/j.ijrobp.2008.12.075. Epub 2009 May 21. PMID 19464819
- [Derived] Lee J, Nguyen NT, Wright J, Yeung KD, Sagar S, Kim DH, Ostapiak O, Doerwald-Munoz L, Whelan T. A phase 2 study of stereotactic body radiation therapy for squamous cell carcinoma of the head and neck (SHINE): a single arm clinical trial protocol. BMC Cancer. 2023 Apr 26;23(1):379. doi: 10.1186/s12885-023-10807-4. PMID 37098494
- See also: Cancer Statistics. National Cancer Institute. — http://www.cancer.gov/